CLINICAL TRIAL: NCT03489733
Title: The Effect of Low Protein, Extensively Hydrolyzed Infant Formula on Allergy Prevention in At-risk Infants up to 1 Year of Age: a Randomized, Double-blind, Controlled Intervention Study and the Long-term Effect on Allergy Prevention of Early Nutrition Given in the First 120 Days of Life in At-risk Infants Until the Child is 6 Years of Age
Brief Title: Prevention of Allergic Diseases in Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HiPP GmbH & Co. Vertrieb KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 508917
Record Dates: First submitted 2018-03-26; First posted 2018-04-05 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Atopic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): Infant Formula with hydrolyzed protein and breast milk until at least 120 days of life
  Interventions: Other: Hydrolyzed Formula
- Control Group (Experimental): Infant Formula with intact protein and breast milk until at least 120 days of life
  Interventions: Other: Control formula
- Breast Fed Group (No Intervention): Exclusively breast ilk until at least 120 days of life

INTERVENTIONS:
Other: Hydrolyzed Formula — Infant formula with extensively hydrolyzed proteins and pre- and probiotics.
  Arms: Intervention Group
Other: Control formula — Infant formula with intact proteins and pre- and probiotics.
  Arms: Control Group

SUMMARY:
A multi-center, prospective, randomized, controlled, doubleblind intervention clinical Trial is performed to proof the efficiency of hydrolyzed infant formula showing a risk reduction of developing an allergy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term-born male and female infants (gestational Age ≥37+0, singleton birth)
* Birth weight ≥ 2500 g and ≤ 4500 g
* Age at enrollment: ≤ 56 days of life
* At risk of developing atopic diseases
* Free of atopy symptoms at Screening and at any time before randomization
* Feeding regimen at any time before Screening (V1) and Baseline (V2, infants who will receive Interventional Product (IP)): no infant formula feeding and solid foods allowed (in order to exclude prior sensitization) except amino acid formula (e.g. Neocate Infant), maltodextrin or glucose solution/gel; breastfeeding allowed
* Subject's parents/caregivers willing to comply with the feeding regimen during the intervention period. Subject's parents/caregivers will decide which feeding regimen will be used (IP or breast milk):

  * IP regimen (intervention or control group): only IP and breast milk until at least 120 days of life
  * breastfeeding regimen (reference group): exclusively breast milk until at least 120 days of life.
  * No other infant formulas or solid foods are allowed.
* Written informed consent.

Exclusion Criteria:

* Multiple births
* Premature delivery (gestational age ≤ 36+6)
* Neonatal illnesses that might have an impact on allergy development (based on Investigator's decision)
* Significant congenital abnormalities
* Participation in another clinical study with an IP or study method that would influence the outcome of this study
* Reason to presume that the subject's parents/caregivers are unable to meet study plan requirements.

Max Age: 56 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1170 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of atopic dermatitis | 1 year
  Presence of atopic dermatitis on physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Beyer, Prof Dr med, Principal Investigator — Charite University, Berlin, Germany
Locations (14):
- Second specialized obstetric and gynecological hospital for active treatment Sheinovo EAD, Sofia, Bulgaria
- Nemocnice Strakonice, a.s., Strakonice, Czechia
- Suomen Terveystalo Oy, Tampere, Finland
- CHU Estaing, Clermont-Ferrand, France
- Germany (5):
  - Charité Universitätsmedizin Berlin, Berlin
  - Klinik für Kinder- und Jugendmedizin der Ruhruniversität Bochum im St. Josef Hospital, Bochum
  - Studienambulanz der pädiatrische Pneumologie und AllergologieKlinik für Kinder- und Jugendmedizin (KKJM), Frankfurt
  - Klinik für Kinder und Jugendmedizin, Hamm
  - Klinik für Kinder- und Jugendmedizin Marienhospital gGmbH Wesel, Wesel
- Unità Allergologia-Unità Allergologia-, Roma, Italy
- Instytut Mikroekologii, Poznan, Poland
- Hospital braga, Braga, Portugal
- Clinical Hospital Center "Dr Dragisa Misovic-Dedinje", Belgrade, Serbia
- Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, Spain